CLINICAL TRIAL: NCT06579131
Title: The Physiotherapeutic Perspective on
Brief Title: Seating Posture and Its Relation to Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, AYŞE KAYALI VATANSEVER, Assistant Professor, Izmir Bakircay University
Other Study IDs: 1111-BAO
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Posture; Myositis; Sitting Position
MeSH Terms: conditions — Myositis | interventions — Sitting Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: sitting position — The participants' seating positions will be assessed, and evaluations will be made based on this.

SUMMARY:
A study has been designed to evaluate pain levels experienced by subjects in relation to different sitting postures. The objective is to investigate how various ergonomic sitting positions affect pain intensity, by systematically assessing pain across a range of sitting postures to identify significant differences and correlations.

DETAILED DESCRIPTION:
A study has been designed to evaluate the pain levels experienced by subjects in relation to different sitting postures. The primary objective of this research is to investigate how various ergonomic sitting positions impact the intensity of pain reported by individuals. This will involve systematically assessing pain levels across a range of sitting postures to determine any significant differences and correlations. The findings are expected to provide insights into the relationship between sitting posture and pain, potentially guiding recommendations for ergonomic improvements.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 65, Not having undergone any surgery affecting spinal posture in the last two years

Exclusion Criteria:

* • Psikiyatrik hastalık tanısı olması ya da tedavi alıyor olması Omurganın duruşunun etkilenmesine sebep olabilecek nörolojik, romatizmal, ortopedik hastalık tanısı almış olmak

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Volunteers from the healthy population
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
pain assessment | 1 year

IPD SHARING:
Plan to Share IPD: Undecided